CLINICAL TRIAL: NCT06009185
Title: An Open-label, Multicentre Study to Evaluate the Safety and Efficacy of Zamicastat as Adjunctive Therapy in Long-term Treatment of Pulmonary Arterial Hypertension (PAH) Disease
Brief Title: Safety and Efficacy of BIA 5-1058 in PAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-202; 2018-002796-18 (EudraCT Number)
Record Dates: First submitted 2023-07-17; First posted 2023-08-24 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; BIA 5-1058; Zamicastat; Bial; Bial - Portela & Ca, S.A.; dopamine ß-hydroxylase (DßH) inhibitor; vascular obstruction; pulmonary arteries; right-heart catheterisation (RHC); idiopathic; rare lung disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTD < 200 mg zamicastat (Experimental): Tablets for oral administration under fed conditions. Zamicastat has to be taken in the morning after breakfast. Each patient will continue treatment with the individual highest tolerated dose (HTD) he/she was taking at MPV3 of the study BIA-51058-201 and will take this dose until visit V5.
  Interventions: Drug: Oral zamicastat
- HTD 200 mg zamicastat (Experimental): Tablets for oral administration under fed conditions containing 100 mg of zamicastat (two tablets of 100 mg). Zamicastat has to be taken in the morning after breakfast. Each patient will continue treatment with the individual highest tolerated dose (HTD) he/she was taking at MPV3 of the study BIA-51058-201 and will take this dose until visit V5.
  Interventions: Drug: Oral zamicastat

INTERVENTIONS:
Drug: Oral zamicastat — Tablets for oral administration under fed conditions containing 100 mg of zamicastat. Zamicastat has to be taken in the morning after breakfast.

SUMMARY:
This study aims to assess the safety and tolerability of the individual highest tolerated zamicastat doses, achieved in the study BIA-51058-201, during long-term treatment in Pulmonary Arterial Hypertension (PAH) disease.

DETAILED DESCRIPTION:
This is an extension study with Pulmonary Arterial Hypertension (PAH) patients who are under treatment with zamicastat as adjunctive therapy in the study BIA-51058-201.

For patients participating in this extension study, visit "Maintenance Period Visit 3" (MPV3) of the study BIA-51058-201 will also be the first visit (V1) of this extension study (BIA-51058-202). Their treatment with zamicastat will be continued at their individual highest tolerated dose (HTD) for an additional 12 weeks (50 mg, 100 mg, 150 mg or 200 mg).

Further visits will be performed 20 ±3 days (V2, telephone), 41 ±3 days (V3, on-site), 62 ±3 days (V4, telephone) and 83 ±3 days (V5, on-site) after V1. At V5, patients will have the opportunity to continue treatment with zamicastat in a compassionate use program. Patients who will not participate in this compassionate use program will come to the following follow-up visit(s):

* Follow-up (FU) down-titration (telephone, 14 ±2 days after V5); only applicable in patients taking 150 mg or 200 mg zamicastat
* FU visit (on-site, 14 ±2 days after last investigational medicinal product (IMP) intake).

The data and safety monitoring board (DSMB) will periodically review the safety data and will issue a recommendation if the study can be continued as planned.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the extension study, patients had to fulfil all of the following criteria at visit V1 (Day 1, start of the extension study):

* Have performed MPV3 of the preceding study BIA-51058-201.
* Able to comprehend and willing to sign an informed consent form (ICF).
* For women: Agreed not to donate ova from the time of informed consent until 30 days after the last IMP intake.
* For men: Agreed not to donate sperm from the time of informed consent until 90 days after the last IMP intake

Exclusion Criteria:

Patients were to be excluded for any one of the following reasons:

* Significant non-compliance with the protocol during the preceding study BIA-51058-201 which may have an impact on this extension study.
* WHO functional class IV as judged by the investigator (reference 1)
* Two or more consecutive measurements of systolic blood pressure (SBP) < 95 mmHg or diastolic blood pressure (DBP) < 50 mmHg measured at visit V1.
* Uncontrolled diabetes mellitus with HbA1c ≥ 8.5% within the last three months or at visit V1.
* Occurrence of an AE during the preceding study which is judged by the investigator as contraindicative to further participation in the extension study.
* Any disease known to cause pulmonary hypertension other than PAH WHO Group 1.
* Obstructive lung disease: Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) < 60% and FEV1 < 60% of predicted value after bronchodilator administration, as demonstrated and documented by previous spirometry data which, in the opinion of the investigator, represent the clinical state of the patient at the time of visit V1.
* Restrictive lung disease: Total Lung Capacity (TLC) < 70% of predicted value, as demonstrated and documented by previous spirometry data which, in the opinion of the investigator, represent the clinical state of the patient at the time of visit V1.
* History of moderate to severe hepatic impairment (Child-Pugh B and C).
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 (measured at Maintenance period visit 1 (MPV1) of study BIA-51058-201).
* Use of the following prohibited medication or treatments during study participation: calcium channel blockers (CCBs) if used for the treatment of PAH in vasoreactive patients; drugs containing a catechol group that is metabolised by DβH (e.g. rimiterole, isoprenaline, dopamine, dopexamine or dobutamide) or α- and/or β-blockers.
* Presence of any other significant or progressive/unstable medical condition that, in the opinion of the investigator, would compromise evaluation of the study treatment or may jeopardise the patient's safety, compliance or adherence to protocol requirements.
* For women: Pregnancy or breast-feeding. Women of childbearing potential unable or unwilling to undergo pregnancy tests and practice highly effective contraceptive measures in combination with a barrier method e.g. condom (without spermicidal foam/gel/film/cream/suppository or fat- or oil-containing lubricants), occlusive cap (diaphragm or cervical/vault caps) with spermicidal gel/film/cream /suppository from the time of informed consent until 30 days after the last IMP intake. Highly effective methods for women are surgical intervention (e.g. bilateral tubal occlusion), non-hormonal implantable intrauterine device, true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the patient) and vasectomised partner (provided that the partner is the sole sexual partner of the patient and the partner has received medical assessment of the surgical success). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), hormonal contraceptives and withdrawal are not acceptable methods of contraception.
* For men: Male patients who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved acceptable contraceptive measure from the time of informed consent until 90 days after the last IMP intake. The following methods are acceptable methods of contraception: partner's use of combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); partner's use of progestogen-only hormonal contraception (oral, injectable/implantable, intrauterine hormone-releasing system); partner's use of implantable intrauterine device; surgical sterilisation (for example, vasectomy or bilateral tubal occlusion).
* Concurrent participation in any other drug investigational study except BIA-51058-201.
* Vulnerable patients according to Section 1.61 of the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guideline for Good Clinical Practice E6.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 12 weeks
  The number of participants with AEs will be presented. An AE is any untoward medical occurrence in a patient to whom a medicinal product is administered and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease occurring during the course of the study.
Clinically relevant changes in laboratory parameters: coagulation | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  Based on coagulation analysis measurements of prothrombin time test (international normalized ratio). The prothrombin time (PT) test measures how long it takes for a clot to form in a blood sample. The International Normalized Ratio is a type of calculation based on PT test results. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Incidence of clinically relevant changes (abnormalities) in laboratory parameters: biochemistry | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  Based on biochemistry analysis measurements (mmol/L) of Sodium, Potassium, Chloride, Calcium, Phosphate . Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Incidence of clinically relevant changes (abnormalities) in laboratory parameters: haematology | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  Based on haematology analysis measurement haemoglobin (g/dL). Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Clinically relevant changes in laboratory parameters: urinalysis | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  Based on urinalysis analysis measurements of the potential of hydrogen (pH). The pH scale is used to determine the degree of acidity of a substance. The basic pH scale extends from 0 (strong acid) to 7 (neutral, pure water) to 14 (strong caustic). Urine has the widest range of pH compared to other bodily fluids. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Clinically relevant changes in laboratory parameters: arterial blood gas | From baseline to week 12, and from day -1 to week 12
  Based on arterial blood gas analysis measurements of Fraction of Inspired Oxygen (%). The fraction of inspired oxygen is the concentration or percentage of oxygen in the air that is inhaled by a person. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Clinically relevant changes in vital signs: blood pressure | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  Systolic and diastolic blood pressure (mmHg) will be measured after the patient has rested for at least 5 minutes in supine position (first measurement) and at least one minute after the first measurement (second measurement). Afterwards, systolic and diastolic blood pressure will be measured again in standing position after the patient has been standing for at least 3 minutes (third measurement). Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Clinically relevant changes in vital signs: pulse rate | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  Pulse rate (bpm) will be measured after the patient has rested for at least 5 minutes in supine position (first measurement) and at least one minute after the first measurement (second measurement). Afterwards, vital signs will be measured again in standing position after the patient has been standing for at least 3 minutes (third measurement). Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Clinically relevant changes in electrocardiogram ECG parameter QT interval | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  QT interval measures the time (msec) it takes the heart muscle to contract and then recover.
  Baseline values will be obtained from V1/A1 of study BIA-51058-201. At Baseline of BIA-51058-201 study and week 12, triplicate 12-lead ECG will be recorded before IMP intake as well as 4 and 8 hours after IMP intake.
Clinically relevant changes in electrocardiogram ECG parameter QRS duration | From baseline to week 6 and week 12, and from day -1 to week 6 and week 12
  The QRS duration measures the time (msec) required for a stimulus to spread through the heart ventricles (ventricular depolarization).
  Baseline values will be obtained from V1/A1 of study BIA-51058-201. At Baseline of BIA-51058-201 study and week 12, triplicate 12-lead ECG will be recorded before IMP intake as well as 4 and 8 hours after IMP intake.

SECONDARY OUTCOMES:
Changes in haemodynamic parameters: pulmonary vascular resistance (PVR) | From Baseline to week 12, and from Day -1 to week 12
  Pulmonary vascular resistance (measured in dyn*s/cm^5) is determined by right heart catheterization to be performed before IMP intake. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in haemodynamic parameters: right atrial pressure (RAP) | From Baseline to week 12, and from Day -1 to week 12
  Right atrial pressure (RAP), measured in mmHg units, is a robust predictor of the pulmonary hypertension severity. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in haemodynamic parameters: mean pulmonary artery pressure (mPAP) | From Baseline to week 12, and from Day -1 to week 12
  Haemodynamic parameter mean pulmonary artery pressure (mPAP) is measured in mmHg units. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in haemodynamic parameters: Cardiac index (CI) | From Baseline to week 12, and from Day -1 to week 12
  Cardiac index (CI) is a haemodynamic parameter that relates the cardiac output from left ventricle in one minute to body surface area, thus relating heart performance to the size of the individual. The unit of measurement is liters per minute per square meter (L/min/m2). Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in haemodynamic parameters: mixed venous oxygen saturation (SvO2) | From Baseline to week 12, and from Day -1 to week 12
  SvO2 is the percentage (%) of oxygen bound to hemoglobin in blood returning to the right side of the heart. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in the New York Heart Association / World Health Organization (NYHA/WHO) functional class | From baseline to week 6 and week 12, and from day -1 to week 12
  The NYHA/WHO Classification system is a tool that classifies patients with heart failure into one of four classes according to their degree of symptoms at rest and with activity: Class I, patients with pulmonary hypertension but without resulting limitation of physical activity; Class II, patients with pulmonary hypertension resulting in a slight limitation of physical activity; Class III, patients with pulmonary hypertension resulting in marked limitation of physical activity; Class IV: patients with pulmonary hypertension with inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnoea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in the 6-minute walk test (6-MWT): Distance Covered | From baseline to week 6 and week 12, and from day -1 to week 12
  The 6-MWT is a self-paced test of walking capacity used to assess aerobic capacity and endurance. It plays a key role in evaluation functional exercise capacity, assessing prognosis and evaluating response to treatment across a wide range of respiratory diseases. The distance covered (m) over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in Biomarker N-terminal pro brain natriuretic peptide (NT-proBNP) | From baseline to week 6 and week 12, and from day -1 to week 12
  NT-proBNP levels in the blood are used for screening, diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure, as this marker is typically higher in patients with worse outcome. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in echocardiogram parameters | From baseline to week 6 and week 12, and from day -1 to week 12
  Parameters used include tricuspid regurgitation, right ventricular contractility, pericardial effusion, right atrial end-systolic area, right ventricular end-diastolic area. Tricuspid regurgitation is a type of heart valve disease in which the valve between the two right heart chambers doesn't close properly. As a result, blood leaks backward into the upper right chamber.
  In was classified as absent, mild, moderate or severe. The right ventricle is the major determinant of functional state and prognosis in PAH. It was measured via tricuspid annular plane systolic excursion (TAPSE). A TAPSE value < 17 mm is considered to indicate right ventricular dysfunction. A pericardial effusion refers to the accumulation of fluid in the pericardial sac surrounding the heart. It was classified as absent (low risk), traces or present (high risk). Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Changes in Quality of life 36-item Short Form Health Survey version 2 (SF-36v2) | From baseline to week 6 and week 12, and from day -1 to week 12
  The SF-36v2 asks 36 questions (items) to measure the functional health and well-being from the patient's point of view. All 36 questions, except question 2 are used to score the 8 health domains. A total score was calculated for each health domain by taking the sum of the corresponding responses and rescaling it to a range of 0 to 100, where 100 represented the best possible result. Baseline values will be obtained from V1/A1 of study BIA-51058-201.
Minimum Plasma Concentration (Cmin) of zamicastat and its metabolites (BIA 5-961 and BIA 5-453) | Day -1, week 6 and week 12
  The pharmacokinetic (PK) parameter Minimum Plasma Concentration (Cmin) for zamicastat and its metabolites will be derived at the end of the dosing interval. Cmin will be measured in ng/mL units. Blood samples will be obtained prior to IMP intake.
Changes in plasma of dopamine ß-hydroxylase (DβH) activity | From baseline to week 6 and week 12, and from day -1 to week 12
  The assessment of plasma DβH activity (% inhibition) was performed centrally. Blood sampling for the assessment of plasma DβH activity was to be performed together with the PK blood sampling. Blood samples were to be taken prior to IMP intake. Baseline values will be obtained from V1/A1 of study BIA-51058-201. Day -1 visit
Catecholamine (norepinephrine and dopamine) levels urinary pharmacodynamic change from baseline: changes in 24-hour | From baseline to week 6 and week 12, and from day -1 to week 12
  24-hour urine collection was to be started on the day before the respective visit. Results for norepinephrine and dopamine are given in nmol per 24 hours (nmol/24hr).

CONTACTS AND LOCATIONS:
Locations (11):
- Ordensklinikum Linz Elisabethinen, Interne 2 - Kardiologie, Angiologie & Interne Intensivmedizin Fadingerstraße 1, Linz, Austria
- Universitätsklinikum Carl Gustav Carus Dresden, Medizinische Klinik und Poliklinik I, Pneumologie Fetscherstraße 74, Dresden, Germany
- Italy (2):
  - ASST di Monza-Ospedale San Gerardo -Dipartimento di Pneumologia via Pergolesi 33, Monza
  - AOU di Roma-Policlinico Umberto I-Unità Dipartimentale Malattie del Circolo Polmonare Viale del Policlinico 155, Roma
- Centro Hospitalar Lisboa Norte, E.P.E. - Hospital Pulido Valente Consulta Externa de Hipertensão Pulmonar Alameda das Linhas de Torres, 117, Lisbon, Portugal
- Spain (4):
  - Hospital Clinic de Barcelona Calle Villarroel, 170, Barcelona
  - Hospital Universitario "12 de Octubre" Avda. de Córdoba, s/n, Madrid
  - Complejo Asistencial Universitario de Salamanca Pº. San Vicente, 58, Salamanca
  - Hospital Universitario Marques de Valdecilla Avenida Valdecilla, 25, Santander
- United Kingdom (2):
  - Golden Jubilee National Hospital Golden Jubilee National Hospital Agamemnon St, Scottish Pulmonary Vascular Unit Golden Jubilee National Hospital, Clydebank
  - Royal Free Hospital Pond Street, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355